CLINICAL TRIAL: NCT02459652
Title: Phase II Study of Neoadjuvant S-1 and Concurrent Radiotherapy for Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant S-1 and Concurrent Radiotherapy for Borderline Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Adjuvant Study Group of Pancreatic Cancer (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Pharma Valley Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JASPAC 05
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Cancer
Keywords: Borderline Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); Radiotherapy

ARMS (1):
- Neoadjuvant S-1/RT (Experimental): This is a single arm prospective study. All eligible subjects will receive neoadjuvant S-1 and concurrent radiation followed by surgical resection. Subjects may receive adjuvant chemotherapy after surgical resection at the clinical discretion of the medical oncologists.
  Interventions: Drug: S-1; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: S-1 — S-1 is administered orally at a dose of 40 mg/m2 twice daily on the day of irradiation (Monday through Friday) during radiation therapy.
Radiation: Radiation Therapy — Radiation therapy is delivered with >6-megavolts (MV) photons, using a multiple field technique. A total dose of 50.4 Gy is delivered in 28 fractions over 5.5 weeks.

SUMMARY:
Multicenter Prospective Phase II Study for Neoadjuvant S-1 and Concurrent Radiotherapy for Borderline Resectable Pancreatic Cancer

RATIONALE: Borderline resectable pancreatic cancer is frequently related to a positive surgical margin and has a poor prognosis after resection. Neoadjuvant chemoradiation with intensive local effect may lead to substantial local control and prolongation of survival in borderline resectable pancreatic cancer.

PURPOSE: This phase II trial assess efficacy and safety of neoadjuvant S-1 and concurrent radiotherapy for borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
S-1: S-1 is an oral fluorinated pyrimidine agent which contains tegafur (FT, a prodrug of 5-FU), 5-chloro-2,4-dihydropyrimidine (CHDP) and potassium oxonate (Oxo) effective for gastric and various other types of cancers. S-1 is also active for pancreatic cancer: S-1 demonstrated non-inferiority to gemcitabine in overall survival for metastatic or locally advanced pancreatic cancer (LAPC).

S-1 and Concurrent radiotherapy: S-1 therapy with concurrent radiation therapy (RT) had favorable activity with overall tumor response rate of 37%, as well as mild toxicity in patients with LAPC. The median survival time and the 2-year survival rate for LAPC patients treated by S-1/RT were 16.2 months and 26% respectively.

Definition of Borderline Resectable Pancreatic Cancer:(1) Reconstructible bilateral impingement of superior mesenteric vein or portal vein; (2) Tumor contact with the superior mesenteric artery (SMA) of </= 180 degrees ; (3) Tumor contact with the common hepatic artery of </= 180 degrees (at the root of the gastroduodenal artery); and (4) Tumor contact with the celiac axis of </= 180 degrees.

Tumor with portal vein tumor thrombus and tumor contact with the second or further jejunal SMA branch are considered as unresectable. Tumor which is contact with the common hepatic artery or celiac axis but can be resected by distal pancreatectomy with en bloc celiac axis resection, is not included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof of pancreatic ductal carcinoma or adenosquamous carcinoma is required prior to study entry.
* Disease assessment by Multi Detector-row Computed Tomography (MDCT) scan within 2 weeks of study entry
* Borderline resectable pancreatic cancer
* No evidence of metastatic disease as determined by chest CT scan, and abdominal CT scan and laparoscopy. Paraaortic lymph node metastasis is considered as metastatic.
* Age >/=20 years old, </=75 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* No prior chemotherapy or radiotherapy for pancreatic cancer
* A square 10 x 10 cm radiation field could encompass all pancreatic lesions and lymph node metastases
* Adequate oral intake
* Appropriate biliary drainage for obstructive jaundice
* Lab Values:

  * hemoglobin concentration >/= 9.0 g/dL
  * leukocyte count >/= 3,000/mm3
  * platelet count >/= 100,000/mm3
  * serum total bilirubin </= 2.0 mg dL, or </=3.0 mg/dL with biliary drainage
  * Aspartate Transaminase (AST) and Alanine Transaminase (ALT) </= 100 U/L, or </= 150 U/L with biliary drainage
  * serum albumin >/= 3.0 g/dl
  * serum creatinine </= 1.2 mg dL
  * Creatinine clearance >/= 50 ml/min
* Written informed consent

Exclusion Criteria:

* Tumor invasion to the alimentary tract determined by abdominal CT scan or endoscopic examination
* Prior chemotherapy using fluoropyrimidine
* Prior radiation therapy to the abdomen
* Watery diarrhea
* Concurrent phenytoin, warfarin potassium, or flucytosine treatment
* Presence of contrast medium allergy
* Pulmonary fibrosis or interstitial pneumonia
* Pleural effusion or ascites
* Active infection
* Uncontrolled diabetes mellitus (FBS >/= 200mg/dL or HbA1c >/= 10.0)
* Active concomitant malignancy
* Active gastroduodenal ulcer
* Severe complications such as cardiac or renal disease
* Regular administration of systemic corticosteroid
* Psychiatric disorder
* History of drug hypersensitivity
* Pregnant and lactating women and women of childbearing age who were not using effective contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-12-28 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | Up to 4 years
  R0 resection rate of all patients enrolled in the study

SECONDARY OUTCOMES:
Overall survival | up to 6 years
Disease-free survival | up to 6 years
Response rate after neoadjuvant chemoradiation | Up to 4 years
  All responses will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 within 4 weeks after completion of neoadjuvant therapy.
Pathological response rate | Up to 4 years
  Evaluation of the pathological response of the primary tumor was performed using a classification by Evans et al.
2-year survival rate | up to 6 years
Surgical morbidity rates | With in 90 days
  Both Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and Clavien-Dindo Classification will be used for all morbidity assessments.
Acute and late toxicity rates | With in 6 months
  All toxicities will be measured by CTCAE version 4.0.
R0 resection rate in borderline resectable pancreatic cancer | Up to 4 years
  Diagnosis of borderline resectable pancreatic cancer will be fixed by Diagnostic Radiology Central Review.

CONTACTS AND LOCATIONS:
Overall Officials: Masafumi Ikeda, M.D., Ph.D., Principal Investigator — National Cancer Center Hospital East, Department of Hepatobiliary Pancreatic Oncology; Katsuhiko Uesaka, M.D., Ph.D., Study Chair — Shizuoka Cancer Center Hospital
Locations (22):
- Japan (22):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Asahikawa Medical University, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Hospital Organization Osaka National Hospital, Chuo-ku, Osaka
  - Saitama Cancer Center, Kita-adachigun Inamachi, Saitama
  - Seirei Mikatahara General Hospital, Hamamatsu, Shizuoka
  - Shizuoka Cancer Center, Suntohgun, Nagaizumityo, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Tokyo Women's Medical University Hospital, Shinjuku, Tokyo
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyusyu Cancer Center, Fukuoka
  - Yamagata University Hospital, Yamagata

REFERENCES:
- [Background] Takahashi S, Ohno I, Ikeda M, Kobayashi T, Akimoto T, Kojima M, Konishi M, Uesaka K. Neoadjuvant S-1 with concurrent radiotherapy followed by surgery for borderline resectable pancreatic cancer: study protocol for an open-label, multicentre, prospective phase II trial (JASPAC05). BMJ Open. 2017 Oct 22;7(10):e018445. doi: 10.1136/bmjopen-2017-018445. PMID 29061632
- [Background] Takahashi S, Ohno I, Ikeda M, Konishi M, Kobayashi T, Akimoto T, Kojima M, Morinaga S, Toyama H, Shimizu Y, Miyamoto A, Tomikawa M, Takakura N, Takayama W, Hirano S, Otsubo T, Nagino M, Kimura W, Sugimachi K, Uesaka K. Neoadjuvant S-1 With Concurrent Radiotherapy Followed by Surgery for Borderline Resectable Pancreatic Cancer: A Phase II Open-label Multicenter Prospective Trial (JASPAC05). Ann Surg. 2022 Nov 1;276(5):e510-e517. doi: 10.1097/SLA.0000000000004535. Epub 2020 Oct 15. PMID 33065644